CLINICAL TRIAL: NCT04447443
Title: Impact of Dietary Fiber as Prebiotics on Chemotherapy-related Diarrhea in Patients With Gastrointestinal Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: discontinued prematurely by sponsor for strategic reasons
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Cancer Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Jinhua Municipal Central Hospital (Other); Quzhou Kecheng People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-111
Record Dates: First submitted 2020-06-17; First posted 2020-06-25 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Chemotherapy-related Diarrhea
MeSH Terms: interventions — Loperamide; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic Fiber (Experimental)
  Interventions: Dietary Supplement: Prebiotic Fiber Supplement + loperamide hydrochloride capsule
- Maltodextrin (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin + loperamide hydrochloride capsule

INTERVENTIONS:
Dietary Supplement: Prebiotic Fiber Supplement + loperamide hydrochloride capsule — 2-week sequential supplementation with prebiotic fiber supplement (3.5g, twice a day).
  The initial dose of loperamide hydrochloride capsules is 4 mg (2 capsules) followed by 2 mg/4 h if diarrhea persists.
  Arms: Prebiotic Fiber
Dietary Supplement: Maltodextrin + loperamide hydrochloride capsule — 2-week sequential supplementation with placebo of of maltodextrin (3.5g, twice a day).
  The initial dose of loperamide hydrochloride capsules is 4 mg (2 capsules) followed by 2 mg/4 h if diarrhea persists.
  Arms: Maltodextrin

SUMMARY:
This study evaluates longitudinal data associating changes in gut microbiota composition and diversity, defecation, performance status and adverse reactions in response to prebiotic fiber supplementation in patients with gastrointestinal cancer chemotherapy-related diarrhea. 120 adult participants , age 18 to 65 years, will be randomized into one of the two arms. Arm A (intervention group) will receive prebiotic fiber and loperamide hydrochloride capsule(a drug for standard treatment). Arm B will receive maltodextrin placebo and loperamide hydrochloride capsule.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65, be able to comply with the protocol
* Life expectancy greater than 3 months
* Patients with cytologically or histologically confirmed diagnosis of gastrointestinal cancers
* Undergoing chemotherapy, not synchronized with radiotherapy and other anti-tumor treatments
* Chemotherapy-related diarrhea grade 2-4
* Not experience diarrhea before chemotherapy

Exclusion Criteria:

* age<18 or >65
* Patients who cannot eat by mouth for example chewing disorders, difficulty swallowing, intractable vomiting, gastrointestinal obstruction or gastrointestinal tract bleeding
* Other acute or chronic diarrhea or colostomy
* Patients with other severe adverse effects of chemotherapy other than diarrhea
* Patients with severe diseases of heart, kidney, liver and other major organs
* Use of any other drug for promoting intestine movement
* Use of any other drug or dietary supplement for chemotherapy-related diarrhea such as other fiber supplements, probiotics, octreotide
* Allergic to the components of the intervention dietary supplements;
* Pregnancy (positive serum pregnancy test) and lactation
* Any other serious or uncontrolled illness which the investigator think is undesirable for the patient to enter the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Therapeutic effect on the chemotherapy-related grade 2 to 4 diarrhea | 2 weeks
  Numbers of bowel movements per day

SECONDARY OUTCOMES:
onset time | 2 weeks
Adverse events | 2 weeks
  Incidence of mild (e.g. self-resolving), moderate (e.g. those that warrant medical evaluation and treatment) and serious (e.g. those that cannot be resolved by medical treatment) adverse events based on criteria adopted by the National Institute of Health common terminology criteria for adverse events (NIH severity) will be evaluated
Changs in Karnofsky Performance Status | 2 weeks
Gut microbiota changes in response to intervention | Change from baseline in gut microbiota at 1 and 2 weeks ]
  16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Pianhong Zhang, Principal Investigator — Second Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided